CLINICAL TRIAL: NCT03919019
Title: Evaluation of Macular Function and Related Changes in Visual Perception and Retinal Morphology After 6 Months of Use of Oral Supplementation Called MACUPREV, in Patients With Dry Age-related Macular Degeneration (AMD)
Brief Title: Morpho-functional Changes After Oral Supplementation of Antioxidants and Anti-inflammatory Treatment in Age-Related Macular Degeneration.
Acronym: MACUPREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Mariacristina Parravano, Head Retina Unit, Fondazione G.B. Bietti, IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RET 04 2017
Record Dates: First submitted 2019-02-14; First posted 2019-04-18 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Dry AMD
Keywords: oral supplementation; mfERG; OCT

STUDY DESIGN:
Intervention Model Description: monocentric, prospective, double blind randomized six months study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macuprev Group (Experimental): patients taking oral supplementation (Macuprev) 2 capsules per day for 6 months
  Interventions: Other: Macuprev Group
- Placebo Group (Placebo Comparator): patients taking oral placebo 2 capsules per day for 6 months
  Interventions: Other: Placebo Group

INTERVENTIONS:
Other: Macuprev Group — oral supplementation (Macuprev) 2 capsules per day for 6 months
  Arms: Macuprev Group
Other: Placebo Group — oral placebo 2 capsules per day for 6 months
  Arms: Placebo Group

SUMMARY:
In patients with AMD a deterioration of the antioxidant mechanisms of the retina is observed and therefore an increase in the production of free radicals responsible for tissue damage.

The Age-Related Eye Disease Study (AREDS) found that the intake of antioxidants reduces the risk of progression of the disease to an advanced stage (choroidal neovascularization or geographic atrophy ) and reduces the loss of visual acuity.

In this study the investigators want to analyze the functional retinal changes (mfERG) of the macular region, in patients with dry age-related macular degeneration, after the use for 6 months of an oral supplementation based on Ganoderma lucidum (Reishi), Calendula Officinalis, Lutepure-Marigold ( 5% Lutein and 1% Zeaxanthin) Blueberry, Rutin, Alpha-lipoic acid, Bromelain, NAC, Vtiamine C, B9, B12, D3, Selenium, Zinc and Copper.

ELIGIBILITY:
Inclusion Criteria:

* age> 50;
* dry AMD not in therapy with oral supplements or antioxidants
* visual acuity ≥ 20/40
* ability to provide written informed consent and to follow the procedures of the study;

Exclusion Criteria:

* spherical refractive error greater than ±6 diopters
* cylindrical refractive error greater than ±3 dioptres
* opacity of diopter means
* any active or past retinal pathology other than AMD
* history of ocular surgery (<6 months)
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change of Multifocal electroretinogram (mfERG) in patients with dry age-related macular degeneration after 6 months follow up | Functional retinal changes after 6 months follow up
  To evaluate functional retinal changes of the macular region by multifocal electroretinogram in patients with dry age-related macular degeneration after the use for 6 months of an oral supplementation in tablets based on Ganoderma lucidum (Reishi), Calendula Officinalis, Lutepure-Marigold ( 5% Lutein and 1% Zeaxanthin) Blueberry, Rutin, Alpha-lipoic acid, Bromelain, NAC, Vtiamine C, B9, B12, D3, Selenium, Zinc and Copper.
  The researchers analyzed the average response amplitude densities (RAD: nanoV/ degree 2) between the first negative peak, N1 and the first positive peak, P1

SECONDARY OUTCOMES:
To evaluate correlation between mfERG changes (functional activity) and morphological retinal changes (CRT: central retinal thickness and VD: vessel density at the superficial and deep capillary plexa) after 6 months follow up | Morpho-functional retinal relationships after 6 months follow up
  The researchers evaluated the linear relationships between the mfERG (Response Amplitude Density (RAD nanoV/degree2) and OCT/OCTA values (CRT in micron and vessel density in mm3) by Pearson's Test after administration of a oral supplementation (Macuprev)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione G.B.Bietti, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Age-Related Eye Disease Study Research Group; SanGiovanni JP, Chew EY, Clemons TE, Ferris FL 3rd, Gensler G, Lindblad AS, Milton RC, Seddon JM, Sperduto RD. The relationship of dietary carotenoid and vitamin A, E, and C intake with age-related macular degeneration in a case-control study: AREDS Report No. 22. Arch Ophthalmol. 2007 Sep;125(9):1225-32. doi: 10.1001/archopht.125.9.1225. PMID 17846363
- [Background] Parisi V, Tedeschi M, Gallinaro G, Varano M, Saviano S, Piermarocchi S; CARMIS Study Group. Carotenoids and antioxidants in age-related maculopathy italian study: multifocal electroretinogram modifications after 1 year. Ophthalmology. 2008 Feb;115(2):324-333.e2. doi: 10.1016/j.ophtha.2007.05.029. Epub 2007 Aug 22. PMID 17716735
- [Background] Piermarocchi S, Saviano S, Parisi V, Tedeschi M, Panozzo G, Scarpa G, Boschi G, Lo Giudice G; Carmis Study Group. Carotenoids in Age-related Maculopathy Italian Study (CARMIS): two-year results of a randomized study. Eur J Ophthalmol. 2012 Mar-Apr;22(2):216-25. doi: 10.5301/ejo.5000069. PMID 22009916
- [Derived] Parravano M, Tedeschi M, Manca D, Costanzo E, Di Renzo A, Giorno P, Barbano L, Ziccardi L, Varano M, Parisi V. Effects of Macuprev(R) Supplementation in Age-Related Macular Degeneration: A Double-Blind Randomized Morpho-Functional Study Along 6 Months of Follow-Up. Adv Ther. 2019 Sep;36(9):2493-2505. doi: 10.1007/s12325-019-01016-2. Epub 2019 Jun 25. PMID 31243641